CLINICAL TRIAL: NCT05502861
Title: A Pragmatic Trial of an Active Choice Nudge for Generalist or Specialist Palliative Care for Seriously Ill Inpatients: The Palliative Connect Trial
Brief Title: A Pragmatic Trial of an Active Choice Nudge for Generalist or Specialist Palliative Care for Seriously Ill Inpatients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Katherine Courtright, Assistant Professor of Medicine, University of Pennsylvania
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 848497; R01AG073384 (NIH)
Record Dates: First submitted 2022-08-12; First posted 2022-08-16 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Palliative Care
Keywords: Palliative Care, Pragmatic Trial
MeSH Terms: interventions — General Practitioners

STUDY DESIGN:
Intervention Model Description: stepped-wedge cluster (at hospital-level) randomized trial
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The study's intervention is a prognostic-triggered EHR alert to nudge clinicians to provide generalist or specialist PC. The alert notifies the clinician that the patient is likely to benefit from PC, and requires clinicians to actively choose to provide generalist PC themselves, consult PC specialist, or to defer PC. If a clinician chooses to consult specialist PC, a second alert will fire that enables them to easily and quickly place the consult order. The alert will trigger for all patients with moderate or higher 6-month mortality risk on second full hospital day at 8AM.
  Interventions: Behavioral: Generalist + Specialist palliative care
- Control/Usual Care (Active Comparator): During the control phase, patients meeting eligibility criteria will be enrolled for study data collection but there will be no attempt to influence delivery of care. The length of the control phase will differ at each hospital dependent on the sequence in which hospitals are randomly assigned to switch to the intervention phase. All hospitals contribute a minimum of 15 weeks of outcomes data prior to adopting the intervention.
  Interventions: Behavioral: Pre-Intervention phase

INTERVENTIONS:
Behavioral: Generalist + Specialist palliative care — Clinicians are alerted in the EHR to make an active choice whether to provide generalist palliative care themselves, consult PC specialist, or to defer PC at that time.
  Other Names: Active choice generalist palliative care
  Arms: Intervention
Behavioral: Pre-Intervention phase — Patients meeting eligibility criteria will be enrolled for study data collection but there will be no attempt to influence delivery of care.
  Other Names: Usual care
  Arms: Control/Usual Care

SUMMARY:
This stepped-wedge, cluster-randomized pragmatic trial among six hospitals at University of Pennsylvania Health System will test a behavioral intervention embedded within the electronic health record that nudges hospital clinicians to either provide palliative care (PC) themselves (generalist PC) or consult specialists (specialty PC) for inpatients at high risk of death within 6 months. The trial will evaluate the intervention's effect compared to usual care on the primary outcome of hospital-free days through 6 months, and other patient-centered, clinical, and economic outcomes. The trial also includes an embedded mixed methods study to understand clinician and hospital contextual factors that influence the intervention's uptake.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Inpatient or observation admission status at a study hospital
* Predicted 6-month mortality risk moderate (e.g., ≥40%) or higher

Exclusion Criteria:

* Under 18 years of age
* Inpatient primary service: hospice, rehabilitation, obstetrics, psychiatry
* Patients that have died or been discharged before 0800 on hospital day 3 when the mortality risk is generated and enrollment occurs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16000 (Estimated)
Dates: Start 2023-11-13 (Actual); Primary Completion 2026-05-17 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Hospital-free days | 6 months
  Days from enrollment spent alive and not in an acute care hospital through 6 months or death

SECONDARY OUTCOMES:
Goals of Care (GOC) conversation within a discrete GOC note type | up to 6 weeks
  Presence or absence of documented GOC conversation after enrollment detected by natural language programming algorithm or by a discrete GOC note type
Pain scores | up to 6 weeks
  pain level according to standardized scale across hospitals after enrollment
Palliative care consultation note | up to 6 weeks
  Presence or absence of signed inpatient palliative care note after enrollment
Time to palliative care consult | up to 6 weeks
  starts at time of enrollment until receipt of first documented inpatient palliative care consultation note
Change in code status found in chart documentation | up to 6 weeks
  no change, new limitations on life support (e.g., DNAR, DNI) or discontinued limitations on life support
Intensive care unit admission | up to 6 weeks
  admitted to any ICU during hospital encounter
Hospital length of stay | up to 6 weeks
  number of days in hospital staring at enrollment
Hospital all-cause mortality | up to 6 weeks
  death occurred in the hospital or within 1 day of discharge
Hospice enrollment | up to 6 weeks
  yes if new hospice enrollment
Home or clinic palliative care referral | up to 6 weeks
  yes if new home of clinic palliative care order after enrollment
Hospital discharge disposition written in discharge order | up to 6 weeks
  Discharge to home, other acute facility, skilled nursing facility
30-day hospital readmission | 30 days
  readmission within 30 days of discharge
180-day all cause mortality | 180 days
  180 days after enrollment
Hospital total costs | up to 6 weeks
  continuous hospital costs
Future acute care costs | enrollment to 6 months post hospital discharge
  acute care costs over the 6 month follow up period
Goal-concordant care | enrollment to 6 months post hospital discharge
  yes if treatments received over 6 month follow up align with goals documented in the EHR; no if treatments are misaligned with goals, or goals are unclear or undocumented
McGill Quality of Life-Revised | 1 month
  14-item survey instrument; score 0-10; continuous
McGill Quality of Life-Revised | 3 months
  14-item survey instrument; score 0-10; continuous
McGill Quality of Life-Revised | 6 months
  14-item survey instrument; score 0-10; continuous
CMS-MACRA PC Quality | 1 month
  (1) felt heard and understood (4-items); (2) received desired help for pain (3-items); continuous

CONTACTS AND LOCATIONS:
Overall Officials: Katherine R Courtright, MD, MS, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie published results will be made available to other researchers, after deidentification.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available beginning 9 months after publication and up to 36 months following publication. After 36 months the data will be available in our University's data warehouse but without support, except for deposited metadata.
Access Criteria: Proposals for data use will be reviewed by Principal Investigator and independent review boards (such as Institutional Review Board and Data Safety and Monitoring Board). Approved data requestors will need to sign data use agreements to access and use data
URL: http://www.pair.upenn.edu